CLINICAL TRIAL: NCT02803320
Title: Supervised Outdoor -Use Test to Assess the Safety of a Sunscreen Lotion on Sports Users
Brief Title: To Assess the Safety of a Sunscreen Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 18309
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agents
Keywords: Sunscreen active

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPF 50 Y65 110 (Experimental): All subjects received baseline skin evaluation and 1 day of sun exposure.
  Interventions: Drug: SPF 50 Y65 110 (BAY 987516)

INTERVENTIONS:
Drug: SPF 50 Y65 110 (BAY 987516) — Subjects applied the assigned products to all sun-exposed areas of their face and body liberally and evenly, in accordance with instructions. Sun exposure was divided into two periods. Each period consisted of direct sun exposure (out of water; Cycle A) and water exposure (Cycle B). Cycles A and B were repeated two times before study closeout.

SUMMARY:
The objective of this study was to assess the safety and appropriateness of a sunscreen product for use on sport users, under supervised outdoor use conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, 18 to 65 years of age with no medical conditions of the skin as determined by the subjects' dermatological medical history.
* The subject must have Fitzpatrick skin types I to VI.
* During the selection process, potential subjects must agree to restrict their sun exposure activities for at least 5 days immediately preceding participation in the study. Subjects must be willing and physically able to spend approximately 3 continuous hours in the sun, must agree to immerse their entire body under water (including face and hair) at least 2 times during the water activity phase, and must agree to refrain from taking any medications during the study that might alter their response to sun exposure
* Subjects must agree to refrain from alcohol and tobacco use during the course of the study
* Subjects must obey all rules of the test facility
* Subjects must agree to refrain from tanning bed usage and significant non study related sun exposure during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2015-05-31 (Actual)

PRIMARY OUTCOMES:
Dermatologist´s subjective and objective assessments of potential Adverse events | 2 days
  • "product related," • "likely product related," • "unlikely product related, or "not product related.
Final Skin Evaluation | 2 days
  • Score 0 (no response): Normal skin. No visible response or erythema. up to Score 3 (severe response): A well demarcated area of very intense or "beet" red erythema or an area of the skin affected by significant edema, papules, and/or vesicles. Usually symptomatic and may require therapeutic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States